CLINICAL TRIAL: NCT04478877
Title: Establishment and Characterization of Meningioma Patient-derived Organoids
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, George KC Wong, Clinical Professor, Chinese University of Hong Kong
Other Study IDs: GWMO01
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Meningioma
MeSH Terms: conditions — Meningioma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Meningioma tumor sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, meningioma organoids will be established from patients' tissues and the characterization of the organoid will be performed.

DETAILED DESCRIPTION:
Aims and Hypothesis to be tested:

The investigators hypothesized that the derived organoid should have a similar morphological and genetic mutation signatures to the patient primary tissue.

Study period: 1 year for patient recruitment and organoid generation from patient tumor

Study population: 30

Study samples:

Patient's meningioma tumor sample are collected from patients with surgical needs. Sample collected are used for organoid culture. Morphological and genetic characteristics will be compared between the patient tumor sample and the corresponding derived organoids

Primary outcome measures:

Whole exome sequencing data of patient tumor tissue and patients-derived organoids

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (aged >18 years) with meningioma
2. Admission into Prince Wales hospitals neurosurgical services
3. Patients with surgical needs of meningioma removal

Exclusion Criteria:

1. Patients (or next-of-kin as appropriate) refuse to participate into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with meningioma admitted to Prince Wales Hospitals neurosurgical services
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-05-23 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Whole exome sequencing data | 7 days
  DNA extracted from patient tumor tissue and patients-derived organoids will be perform whole exome sequencing for genetic characterization.

SECONDARY OUTCOMES:
Immunostaining | 7 days
  H&E staining and meningioma markers immunostaining

CONTACTS AND LOCATIONS:
Overall Officials: George KC Wong, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Surgery, The Chinese University of Hong Kong, Hong Kong, Hong Kong